CLINICAL TRIAL: NCT07357337
Title: Efficacy of Oral Metformin vs Oral Doxycycline in Treating Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acne Vulgaris on the Face; Acne Vulgaris
Keywords: acne vulgaris; metformin; doxycycline; oral; efficacy
MeSH Terms: conditions — Acne Vulgaris | interventions — Metformin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Group A (Experimental): Group A will receive oral tablet Metformin 500mg twice daily
  Interventions: Drug: oral metformin
- Control Group: Group B (Active Comparator): Group B will receive oral tablet Doxycycline 100mg once daily
  Interventions: Drug: Oral doxycycline

INTERVENTIONS:
Drug: oral metformin — Intervention group will recieve oral tablet Metformin 500mg twice daily
  Arms: Intervention Group: Group A
Drug: Oral doxycycline — Group B will receive oral tablet Doxycycline 100mg once daily
  Arms: Control Group: Group B

SUMMARY:
The goal of the clinical trial is to learn if oral metformin works to treat moderate to severe acne vulgaris.

Investigators will compare this drug to oral doxycycline to see if this drug works to treat acne. All participants will be divided into two groups.

Group A will be given oral Metformin 500 mg to be taken twice daily, while Group B patients will be given oral Doxycycline 100 mg once daily. They will be assessed by the scoring method Total Lesion Count (TLC) and the Global Acne Grading System (GAGS) at each follow-up (i.e., at 0, 8, and 12 weeks). Efficacy will be measured by using the scoring system GAGS, TLC. The final assessment will be done at the 12th-week follow-up.

A total of 68 patients fulfilling the inclusion criteria are enrolled in the study. The efficacy of oral metformin vs oral doxycycline will be measured in all selected patients suffering from acne vulgaris by estimating improvement in the total lesion count (TLC) and the Global Acne Grading (GAGS) assessment score at each follow-up.

DETAILED DESCRIPTION:
Acne vulgaris is a common, long-standing inflammatory condition affecting the pilosebaceous unit. Its main features include follicular plugging and raised inflammatory lesions (papules, pustules, and nodules) and scars (1). Nearly half of the teenagers with acne still experience symptoms as adults. Approximately 70-80% of teenagers have acne (2). In some patients acne can remain as an unremitting disease and cause prolonged psychiatric, psychosocial, and physical consequences.

The development of acne results from a complex series of events occurring within the pilosebaceous unit. (3), encompassing various factors such as pronounced sebum production and modifications in its fatty acid composition. Fluctuations in hormones, increased follicular keratinization (4), and disturbances in both innate and adaptive immune system responses are observed. Together, these complex processes disrupt the normal functioning of the pilosebaceous unit and cause follicular damage; thus, they increase sebum production, fatty acids, and lipids in the skin layer, and they will produce inflammatory and noninflammatory lesions.

Reducing scarring and psychological effects, as well as giving the patient the best possible appearance, are the main objectives of treatment. Treatment goals include preventing follicular hyperkeratosis and preventing the release of fatty acids and sebum, thus decreasing the production of comedones. There are numerous topical and systemic treatment modalities available for acne vulgaris. Commonly prescribed topical therapies for mild acne consist of benzoyl peroxide, retinoids, salicylic acid, azelaic acid, clindamycin, and 5% dapsone (5). Systemic therapeutic approaches for acne that have moderate to severe intensity encompass isotretinoin, tetracycline, doxycycline, metformin, and hormonal therapies. including oral contraceptives and antiandrogens (6). Lasers and light-based therapies can also be used for noninflammatory or mildly inflammatory acne Emerging evidence suggests it is strongly associated with insulin resistance. Increased levels of insulin in the bloodstream, known as hyperinsulinemia, cause an increase in insulin-like growth factor-1 (IGF-1) concentrations accompanied by a decrease in levels of IGFBP3. (insulin-like growth factor binding protein 3 (7). This affects keratinocyte growth and death directly and may cause the release of growth hormone, glucocorticoids, and androgen factors associated with the development of acne.

This novel research will evaluate and compare the therapeutic outcomes of oral metformin and oral doxycycline in the management of moderate to severe acne vulgaris within the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* •Age: 12 years-40 years old

  * Gender: Both Female & Male.
  * Moderate to severe Acne vulgaris (II and III)
  * Able to complete monthly treatment for 12th week
  * Noninflammatory acne

Exclusion Criteria:

* Hypersensitivity or allergic to doxycycline and metformin.
* History of taking systemic medications one month prior.
* Pregnancy and lactation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Total lesion count | change in lesion count over the course of 12 weeks of treatment, with responses assessed at baseline, 4 weeks, and 12 weeks.
Global Acne Grading System (GAGS) | Responses will be assessed at baseline, 4 weeks, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tahreem Alam Buzdar, Principal Investigator — Ghurki Trust Teaching Hospital; Prof. Dr. Haroon Nabi, Study Director — Lahore Medical and Dental College; Dr Aliza Hamadani, Study Chair — Lahore Medical and Dental College; Dr. Ayesha Asad Chattha, Study Chair — Ghurki Trust Teaching Hospital; Dr. Iram Kausar, Study Chair — Ghurki Trust Teaching Hospital
Locations (1):
- Ghurki Trust Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habeshian KA, Cohen BA. Current Issues in the Treatment of Acne Vulgaris. Pediatrics. 2020 May;145(Suppl 2):S225-S230. doi: 10.1542/peds.2019-2056L. PMID 32358215
- [Background] Sadati MS, Yazdanpanah N, Shahriarirad R, Javaheri R, Parvizi MM. Efficacy of metformin vs. doxycycline in treating acne vulgaris: An assessor-blinded, add-on, randomized, controlled clinical trial. J Cosmet Dermatol. 2023 Oct;22(10):2816-2823. doi: 10.1111/jocd.15785. Epub 2023 May 2. PMID 37128834
- [Background] Deng Y, Jiang S, Huang Y, Tan X, Huang Y, Chen L, Xu J, Xiong X, Zhou J, Xu Y. Metformin contributes to the therapeutic effects of acne vulgaris by modifying the gut microbiome. Dermatologic Therapy. 2023;2023(1):9336867.
- [Background] Lee JK, Smith AD. Metformin as an adjunct therapy for the treatment of moderate to severe acne vulgaris. Dermatol Online J. 2017 Nov 15;23(11):13030/qt53m2q13s. PMID 29447630
- [Background] Heng AHS, Chew FT. Systematic review of the epidemiology of acne vulgaris. Sci Rep. 2020 Apr 1;10(1):5754. doi: 10.1038/s41598-020-62715-3. PMID 32238884